CLINICAL TRIAL: NCT01062724
Title: Effect of Two Amino Acid Solutions on Blood Amino Acid Levels and Frequency of Cholestasis in Neonates
Brief Title: Total Parenteral Nutrition Associated Cholestasis (TPNAC) and Plasma Amino Acid Levels in Neonates
Acronym: TPNAC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, María de Lourdes Barbosa Cortés, Associated Researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-785-080
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2016-02

CONDITIONS: Premature Birth
Keywords: Cholestasis; TPN; Neonates; Primene; Trophamine; Methionine; Cysteine; Taurine; Total Parenteral Nutrition
MeSH Terms: conditions — Premature Birth; Cholestasis; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trophamine (No Intervention): This group of neonates will be receive the Trophamine amino acids solution from Pisa laboratories as an active comparator with Primene. The infants in this group will receive, daily intakes (g/kg/d) of parenteral protein, carbohydrate and fat or daily enteral intake (ml/kg/d). Besides, the intake of breast milk or formula will be record, during the first 28 days of total parenteral nutrition.
- Primene 10% from Baxter (Experimental): This group of neonates will be receive the Primene amino acids solution (10 %) from Baxter laboratories as other active comparator with Trophamine. The infants in this group will receive, daily intakes (g/kg/d) of parenteral protein, carbohydrate and fat or daily enteral intake (ml/kg/d). Besides, the intake of breast milk or formula will be record, during the first 28 days of total parenteral nutrition.
  Interventions: Other: Primene 10 % from Baxter

INTERVENTIONS:
Other: Primene 10 % from Baxter — Primene solution will be calculated in g/kg/day and administered in ml/day Active Comparator: Trophamine This group of neonates will be receive the Trophamine amino acid solution from Pisa laboratories and the other arm will be receive a Primene amino acid solution (10 %) from Baxter laboratories. For infants identified, daily intakes (g/kg/d) of parenteral protein, carbohydrate and fat and daily enteral intake (ml/kg/d) of breast milk or formula will be record.
  Other Names: PRIMENE 10%, code IMSS 2512 01 01
  Arms: Primene 10% from Baxter

SUMMARY:
The purpose of this study is to analyze if the infants who received Primene solution, have lower serum levels of methionine and cysteine and higher serum levels of taurine, we also analyze if the infants who received Primene solution develop TPN-associated cholestasis in a smaller proportion than those who received Trophamine solution.

DETAILED DESCRIPTION:
Total parenteral nutrition is an essential component of the care of premature and ill infants. Prolonged parenteral nutrition is associated with complications affecting the hepatobiliary system, such as cholelithiasis, cholestasis, and steatosis. The most common of these is total parenteral nutrition-associated cholestasis (TPNAC), that occurs because of reduced bile flow from the liver into the duodenum. Cholestasis causes liver damage and in some cases, death. Infant and neonate are at particular risk for this complication. The incidence of TPNAC ranges from 7.4 to 84%.

Animal studies have implicated amino acids in the production of cholestasis; whereas studies in human neonates suggest a direct effect of amino acid infusions on the hepatocyte canalicular membrane. An appropriate amino acid solution might compensate for the metabolic immaturity of infants and perhaps reduce total parenteral nutrition associated complications such as cholestasis. Therefore, is important to compare the frequency of cholestasis and blood amino acid concentration during Primene and Trophamine use.

ELIGIBILITY:
Inclusion Criteria:

* Newborns greater than 1500 g who enter the Intensive Care Unit and their pathology requiring total parenteral nutritional support (necrotizing enterocolitis, intestinal atresia, short bowel syndrome).
* Gestational age greater than 30 weeks
* Patients with normal liver function tests for their age, prior to the initiation of total parenteral nutrition.
* Authorization from both parents or legal guardian for recruiting of the child into the study with consent signed form after the purpose and procedures have been explained

Exclusion Criteria:

* Patients with acute renal failure
* Congenital liver disease, end-stage liver disease
* Patients with liver damage secondary to viral or bacterial infection
* Patients with liver damage secondary to drugs

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Blood Amino Acid levels and Frequency of Cholestasis in Neonates | At baseline, day 7, 14, 21 and 28 of the administration of total parenteral nutrition (TPN

CONTACTS AND LOCATIONS:
Overall Officials: Maria de Lourdes Barbosa-Cortés, MSc, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Intensive Care Unit and Nutrition Parenteral Department, Pediatric Hospital , Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765